CLINICAL TRIAL: NCT02458482
Title: Randomized Control Trial of AccuPAP Device Versus Standard Nebulizer Therapy in Acute Asthma Exacerbation in Children
Brief Title: Trial of AccuPAP Device Versus Standard Nebulizer Therapy in Acute Asthma Exacerbation in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The trainee for whom I designed the study did not begin enrollment and has left our institution.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Donald H Arnold, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150070
Record Dates: First submitted 2015-05-22; First posted 2015-06-01 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Asthma
Keywords: Children; Positive Airway Pressure; Nebulizer; Moderate; Acute; AccuPAP
MeSH Terms: conditions — Asthma; Lymphoma, Follicular | interventions — Albuterol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Nebulizer Mask Group (Active Comparator): Patients randomized to this "Control" or "standard therapy" group are to receive current institutional standard therapy for moderate asthma exacerbation which includes 10 mg Albuterol combined with 1.5mg Ipratropium nebulized therapy over one hour.
  Interventions: Drug: Albuterol and Ipratropium Continuous Nebulizer
- AccuPAP Group (Experimental): Patients randomized to this group must also have moderate asthma exacerbation and will use an investigational device called "AccuPAP" to receive three allotments of Albuterol and Ipratropium in nebulized form.
  Interventions: Device: AccuPAP

INTERVENTIONS:
Device: AccuPAP — The AccuPAP device used by participants will give 2.5mg and 0.5mg nebulized Albuterol and Ipratropium over 5 minutes. Inspiratory and expiratory pressures to be set at 6 and 12 cm H20 respectively. This therapy is repeated at 20 and 40 minutes for a total of three AccuPAP treatments.
  Arms: AccuPAP Group
Drug: Albuterol and Ipratropium Continuous Nebulizer — 10mg Albuterol and 1.5mg Ipratropium continuous nebulizer treatment will be administered to a Control group over a one hour period.
  Other Names: Duoneb treatment
  Arms: Standard Nebulizer Mask Group

SUMMARY:
The objective of this randomized control trial is to investigate the efficacy of an adjunct positive airway pressure (PAP) nebulizer device known as "AccuPAP" in the treatment of moderate-severity acute asthma exacerbations in children ages 6 - 17 years in comparison with an institutional standard continuous dual-therapy nebulizer treatment.

The investigators main goal, more specifically, is to determine if the additional positive airway pressure provided by the AccuPAP device when used in treating children with moderate-severity asthma exacerbations provides a more optimal delivery of bronchodilator therapy when compared to institutional standard protocol nebulizer delivery mask which does not employ the use of positive airway pressure in medication delivery. The investigators have determined that the change in a study-validated Acute Asthma Intensity Research Score (AAIRS) which will be considered statistically significant for a patient is 2 points or greater after the first treatment has been completed.

DETAILED DESCRIPTION:
Currently the standard of care for acute asthma exacerbations in children involves immediate administration of an inhaled short acting beta agonist (SABA), most commonly Albuterol, paired with parasympatholytic (Ipratropium) both of which are administered via continuous nebulizer. Additionally, a course of oral or intravenous systemic corticosteroid such as methylprednisolone or decadron are also given to combat acute airway inflammation. Medical providers may also initiate the use of a respiratory support device that can range from supplemental oxygen delivered via nasal cannula (NC) and escalate to the use of Bi-level Positive Airway Pressure (BiPAP) or endotracheal intubation in order to increase delivery of medication to distal airways. Because asthma is the most common chronic disease of childhood, there have been ongoing studies on many fronts which are being undertaken to minimize morbidity, shorten hospitalization duration and more rapidly reduce a patient's level of respiratory distress.

When nebulized medication is delivered to a patient with active bronchospasm it might not be immediately delivered to the smallest bronchioles and terminal airways which are most affected by bronchospasm causing air trapping and poor gas exchange. Current modalities rely on dilation of larger airways first thus allowing medication to diffuse passively to the smaller airways as dilation occurs down the bronchial tree. Medication delivery is passive and dependent upon the progressive relaxation of these larger airways before reaching the smaller airways which is the ultimate goal of nebulized therapies. The critical pressure required for medication to reach these obstructed airways and keep them stented open is higher than in an otherwise healthy individual due to the natural consequences of airway remodeling seen in asthmatics which includes narrowing of the diameter of the airways, increased atelectasis of hypoventilated areas, and overall increased ventilation-perfusion (V/Q) mismatch. The concomitant processes of mucous plugging also commonly seen in asthma further complicates the efficient distribution of these medications in a thoracic cross section. However, application of positive pressure in patients with obstructive airways diseases such as asthma has potential to increase air-trapping, dynamic hyperinflation, and auto-peep and, in turn, aggravate ventilation-perfusion mismatch, all of which has potential to delay clinical improvement. With these considerations, we seek to determine if the physiologic benefit of proposed improved bronchodilator delivery by using added positive airway pressure (ie, active delivery of medication) is of sufficient magnitude to provide overall benefit to patients with acute asthma exacerbation.

The investigators propose to test this hypothesis through the following aim: To conduct a single-blinded (clinical team), randomized clinical trial to determine the efficacy of the AccuPAP device in comparison with the standard nebulizer to decrease acute exacerbation severity measured with the Acute Asthma Intensity Research Score (AAIRS), an objective and validated asthma scoring system, at 0, 1 and 2 hours after initiation of treatment. Secondary outcomes will include Emergency Department (ED) length-of-stay (LOS), general pediatrics floor hospitalization rate, Pediatric Intensive Care Unit (PICU) admission rate, number of patients who do not improve with AccuPAP, and rate of relapse within 24 hours of discharge from the ED. The investigators propose that outcome of the study findings have potential to not only shorten hospital stay duration which is cost efficient but also decrease the burden of the disease process on patient by implementing improved medication delivery strategies.

ELIGIBILITY:
Inclusion Criteria:

* Investigators will enroll children ages 6 - 17 years (inclusive) with a previous diagnosis of asthma who present in an acute exacerbation to the Pediatric Emergency Department.
* Patients will be evaluated using the Acute Asthma Intensity Research Score (AAIRS) which has been validated at Vanderbilt University Medical Center and is currently the standard of care when triaging patients with asthma.
* An included patient's severity of current exacerbation must be qualified using the AAIRS and fall in the moderate category of 7 to 11 points.
* Patients who have received nebulized bronchodilator medications at either a referring facility or at home will be included.
* Patients who present from a referring facility or Primary Care Physician (PCP) and have received systemic corticosteroids (SCS) within one hour of initial AAIRS scoring will also be included.

Exclusion Criteria:

* Exclusion criteria will include the following: other medical conditions contributing to respiratory distress (e.g., pneumonia, cystic fibrosis, anaphylaxis),
* developmental delay or any impedance to following basic AccuPAP use instructions,
* any condition precluding a patient from receiving beta-agonist therapy (ie- predisposition to Supraventricular Tachycardia).
* Patients with a history of spontaneous pneumothorax, recent facial, oral or skull surgery/trauma, history of esophageal surgery, known or suspected tympanic membrane rupture or other middle ear pathology, acute sinusitis, epistaxis, active hemoptysis or nausea will be excluded as these are contraindications for AccuPAP use.
* Patients who have received additional adjunctive therapies beyond repeated SABA and atrovent nebulizers or those who have received SCS greater than 1 hour prior to initial ED evaluation, those who have received intravenous magnesium sulfate infusion, or subcutaneous terbutaline or epinephrine will be excluded.
* Those patients whose parents are require a translator for consent will also be excluded (ie, exclusively Spanish speaking or other non-English speaking families/patients). The justification for this exclusion is that patients with respiratory distress often need rapid initiation of treatment and the delay that may be caused by coordination efforts required in order to obtain a translator for study consent and explanation may delay care for these patients and result in adverse outcomes that may potentially result in harm.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-07 (Estimated); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Change in Acute Asthma Intensity Research Score (AAIRS) | From Initial AAIRS scoring in Triage until the end of hour 1 and 2 of treatment during study enrollment
  A validated asthma scoring system at Vanderbilt University Medical Center used to determine the severity of acute asthma exacerbation

SECONDARY OUTCOMES:
Length of Stay (LOS) | To be determined at the time of patient disposition, usually occuring on average between hours 2 and 4 of emergency department evaluation.
  Time of triage in the Pediatric Emergency Department until Discharge
Rate of Admission to the General Pediatrics Floor | Within 24 hours of study enrollment
  The rate at which patients in both study groups require admission to the general pediatrics hospital floor.
Rate of Admission to the Pediatric Intensive Care Unit (PICU) | Within 24 hours of study enrollment
  The rate at which patients in both study groups require admission to the PICU.
Number of Patients Who Do Not Show Improvement on AccuPAP After the First Hour of Treatment | Within 2 hours of study enrollment
  If a patient appears to worsen on experimental treatment (AccuPAP) by any clinical assessment at any time during their treatment (AAIRS or other clinician assessment), they will automatically be converted to standard nebulizer treatment and dropped from the experimental study group. If a patient's second AAIRS score remains the same as their initial score at 1 hour, they will also be converted to standard nebulizer therapy.
Rate of Relapse | Within 24 Hours of Discharge form the Pediatric Emergency Department
  All patients who return to the Pediatric Emergency Department within 24 hours of discharge with persistent asthma exacerbation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Evan H Allie, MD, Principal Investigator — Pediatric Emergency Medicine Clinical Fellow
Locations (1):
- Vanderbilt University Medical Center Monroe Carell Jr. Childrens Hospital Pediatric Emergency Department, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No